CLINICAL TRIAL: NCT00320346
Title: A Double-Blind, Randomised, Multi-Centre Study to Evaluate the Safety, Tolerability, Immunogenicity and Lot to Lot Consistency of Two Formulations of CSL Limited's Inactivated Prototype Pandemic Influenza Vaccine in a Healthy Adult Population (≤18 Years to ≥64 Years of Age).
Brief Title: Phase II Study of Pandemic Influenza Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Dr Russell Basser, CSL Limited
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CSLCT-PAN-05-18
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2008-11

CONDITIONS: Influenza
Keywords: Pandemic; Influenza; Prevention; Vaccine; Prevention of Pandemic Influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Pandemic Influenza Vaccine

SUMMARY:
The World Health Organisation has warned that an influenza pandemic is inevitable. The avian influenza H5N1 virus strain is the leading candidate to cause the next influenza pandemic. This study will test the safety and immunogenicity of a H5N1 Pandemic Influenza Vaccine in healthy adults. The Study will also assess Lot to Lot consistency of the Pandemic Influenza Vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults

Exclusion Criteria:

* Previous vaccination with an influenza Vaccine containing the H5N1 strain
* History of clinically significant medical conditions
* History of Guillian-Barre Syndrome or active Neurological disease

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400
Dates: Start 2006-07; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Safety and Immunogenicity

SECONDARY OUTCOMES:
Lot to Lot Consistency

CONTACTS AND LOCATIONS:
Overall Officials: Peter Richmond, Dr, Principal Investigator — Princess Margaret Hospital for Children
Locations (3):
- Australia (3):
  - CMAX, a division of IDT Australia, Adelaide, South Australia
  - Murdoch Childrens Research Institute, Melbourne, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia

REFERENCES:
- [Derived] Nolan TM, Richmond PC, Skeljo MV, Pearce G, Hartel G, Formica NT, Hoschler K, Bennet J, Ryan D, Papanaoum K, Basser RL, Zambon MC. Phase I and II randomised trials of the safety and immunogenicity of a prototype adjuvanted inactivated split-virus influenza A (H5N1) vaccine in healthy adults. Vaccine. 2008 Aug 5;26(33):4160-7. doi: 10.1016/j.vaccine.2008.05.077. Epub 2008 Jun 13. PMID 18599164